CLINICAL TRIAL: NCT02608814
Title: Advanced Ultrasound in Pleural Infection
Acronym: AUDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: AUDIO
Record Dates: First submitted 2015-10-21; First posted 2015-11-20 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pleural Infection
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pleural biopsy sampling — 6 - 8 pleural biopsy samples will be taken before the insertion of the chest drain. These samples will be sent to microbiology for examination.
Other: Ultrasound

SUMMARY:
Pleural infection is a potentially serious infection of the fluid normally found around the lung and current evidence suggests its incidence is increasing in both adult and paediatric populations.

Identification of bacterial pathogens causing pleural infection is of paramount importance in the clinical care of patients are currently, only 40% of patients have a laboratory confirmed microbiological diagnosis for their pleural infection. An unclear diagnosis can be due to various reasons such as a small sample volume therefore the aim of the AUDIO study is to ascertain the capacity of pleural biopsies in improving the microbiological yield of pleural infection.

Currently, there are no well validated methods for identifying patients presenting with pleural infection on the basis of initial ultrasound imaging. The AUDIO study will define the role of baseline thoracic ultrasound in predicting the radiographic, clinical and surgical outcomes of patients with pleural infection.

The AUDIO study aims to recruit 50 patients from 2 centres with specific pleural expertise and these patients will be followed up over a 12 month period. Investigators hope that through the information gathered from ultrasound imaging and pleural biopsies, it will aid physicians' clinical and therapeutic decision making when treating patients with pleural infection.

ELIGIBILITY:
Inclusion Criteria:

* A clinical presentation compatible with pleural infection
* A pleural fluid collection that may or (rarely according to clinical judgement) may not require drainage that meets at least one or more of the following criteria:
* Purulent
* Gram stain positive for bacteria
* Bacterial culture positive
* Acidic with a pH <7.2
* Low pleural fluid glucose <3mmol/L (<55mg/dL)
* CT evidence of pleural infection (consolidation of underlying lung with enhancing pleural collection on contrast-enhanced CT)

Exclusion Criteria:

* Age <18 years
* No pleural fluid available for analysis
* Previous pneumonectomy on the side of pleural infection
* Expected survival <3 months due to co-morbid disease
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
To increase microbiological yield. | Positive microbiological results on pleural biopsy at baseline compared with positive microbiological results on pleural fluid.

SECONDARY OUTCOMES:
Radiographic improvement in area of pleural collection measured by the percentage of the ipsilateral hemithorax occupied by effusion on chest radiography. | Day 1 and Day 7
Mortality from pleural infection | 3 and 12 months
Duration of hospital (in patient) stay | From the date of initial hospital admission to the date of discharge assessed up to 2 weeks.
Necessity for surgical fluid drainage documented in case report forms over study completion | 3 and 12 months
Pleural fluid drainage over 7 days | First 7 days of trial involvement

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - North Bristol NHS Trust, Southmead Hospital, Bristol
  - Oxford Respiratory Trials Unit, Churchill Hospital, Oxford